CLINICAL TRIAL: NCT04915105
Title: Personal Precise Treatment on Psoriasis and Psoriatic Arthritis and Investigate the Mechanisms of Biological Agents Induced Systemic Lupus Erythematosus
Brief Title: Personal Precise Treatment on Psoriasis and Psoriatic Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CE20043B
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Dermatologic Disease
Keywords: PSO, PSA, SLE, PBMC
MeSH Terms: conditions — Skin Diseases; Salivary Gland Adenoma, Pleomorphic; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prescreen on psoriasis and psoriatic arthritis treatment (Experimental): Prescreen markers from individual PBMCs and choose proper biologics before starting treatment on psoriasis and psoriatic arthritis patients.
  Interventions: Diagnostic Test: Markers data from PBMCs

INTERVENTIONS:
Diagnostic Test: Markers data from PBMCs — Prescreen markers from patient individual PBMCs treating with streptococcus and different biologics.

SUMMARY:
Part of psoriasis and psoriatic arthritis patients treated with biologics and met primary failure. Therefore, we are going to create a cell based platform to evaluate the treatment effects of different biologics on psoriasis and psoriatic arthritis patients before prescribed by physicians

DETAILED DESCRIPTION:
PBMCs isolated from psoriasis and psoriatic arthritis and incubated with Group A streptococcus and different biologics for 24 hours. Cytokines expression in the culture supernatants will be measured and the data can be reference for physician's prescription.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy control without underline disease such as psoriasis and psoriatic arthritis. 2. Psoriasis been diagnosed for over six months and PASI >10. 3.Psoriatic arthritis been diagnosed for over six months and >1 swallow and tender joints

Exclusion Criteria:

* nil

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
PASI score | 2 weeks to 3 months
  Psoriasis skin condition and severity
swelling joint count and tenderness joint count | 2 weeks to 3 months
  PSA severity

SECONDARY OUTCOMES:
CRP | 3-6 months
  blood test
DLQI | 6 months
  paper to investigate patient life quality

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Yang Yen, MDPhD, Study Chair — Attending Physician

IPD SHARING:
Plan to Share IPD: No